CLINICAL TRIAL: NCT06378164
Title: The Immediate and Sustained Effect of 4-week Combined Volitional and Reactive Step Training in Reducing Falls Risk in Community-Dwelling Older Fallers: a Randomised Controlled Trial
Brief Title: The Effect of Combined Volitional and Reactive Step Training in Reducing Falls Risk in Older Fallers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); Neuroscience Research Australia (Other); The University of New South Wales (Other)
Responsible Party: Principal Investigator, Freddy Man Hin LAM, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0041406
Record Dates: First submitted 2023-11-21; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Older Adults With a History of Falls
Keywords: Falls; Exercise; Randomised Trial; Step Training; Reaction
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined volitional and reactive step training (Experimental)
  Interventions: Behavioral: Exercise
- Non-specific exercise group (Placebo Comparator)
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Exercise — For the combined step training group, the participants will receive training on both volitional and reactive stepping. The training will last for 1 hours per session, 2 session per week for 4 weeks.
  Arms: Combined volitional and reactive step training
Behavioral: Active Control — An active control group will be used to minimise the placebo and history effect. The group will also receive a 4-week programme with the frequency and duration of the training and the instructor-to-participant ratio that match the combined step training group. During training, they will perform exercises not specific to reducing fall risk.
  Arms: Non-specific exercise group

SUMMARY:
To examine the immediate and sustained effect of a 4-week combined volitional and reactive step training on fall risks in community-dwelling older fallers.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* Able to walk for 1 minute under supervision without walking aids
* Have a history of falling in the past year

Exclusion Criteria:

* Cognitive impairment (i.e., scores below the age and education-specific cut-off of 7th percentile in the 5-minute Montreal cognitive assessment)
* Blindness
* Neurological conditions (e.g., stroke, Parkinson's disease)
* Other serious illnesses that preclude participation in exercise training

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Choice Stepping Reaction Times | (i) baseline, (ii) immediately post-intervention, (iii) 3-months post-intervention and (iv) 6-months post-intervention
  To assess volitional stepping performance
Spring Scale Test | (i) baseline, (ii) immediately post-intervention, (iii) 3-months post-intervention and (iv) 6-months post-intervention
  To assess reactive stepping performance

SECONDARY OUTCOMES:
Mini Balance Evaluation System Test | (i) baseline, (ii) immediately post-intervention, (iii) 3-months post-intervention and (iv) 6-months post-intervention
Motor Control Test | (i) baseline, (ii) immediately post-intervention, (iii) 3-months post-intervention and (iv) 6-months post-intervention
Falls Efficacy Scale - International | (i) baseline, (ii) immediately post-intervention, (iii) 3-months post-intervention and (iv) 6-months post-intervention
Trail-Making Test | (i) baseline, (ii) immediately post-intervention, (iii) 3-months post-intervention and (iv) 6-months post-intervention
Programme Adherence | From start to six months after the end of training
  The attendance of the exercise class will be recorded.
Prospective Falls | From start to 12 months after the intervention ends
  Fall incidence and details on fall will be recorded using a fall diary and monthly follow-up.
Adverse Events | From start to six months after the end of training
  Adverse events happened during the intervention will be recorded descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Man Hin LAM, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study data can be provided via contacting the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From Dec 2026 onward
Access Criteria: By contacting the Principal Investigator (Dr Freddy Lam): Freddy-mh.lam@polyu.edu.hk